CLINICAL TRIAL: NCT01328067
Title: A Randomized Study to Evaluate the Safety and Effectiveness of MRgFUS Procedure Compared With Myomectomy for the Treatment of Uterine Fibroids
Brief Title: Study to Evaluate the Safety and Effectiveness of MRgFUS Compared With Myomectomy for the Treatment of Uterine Fibroids
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF034
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Uterine Fibroids; Bleeding; Pelvic Pain
Keywords: MRgFus; Uterine Fibroids; Pelvic Pain; Quality of Life; Symptomatic Uterine Fibroids
MeSH Terms: conditions — Leiomyoma; Hemorrhage; Pelvic Pain | interventions — Uterine Myomectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): MR guided Focused Ultrasound
  Interventions: Device: Exablate 2100
- Surgery (Active Comparator): Myomectomy
  Interventions: Procedure: Myomectomy

INTERVENTIONS:
Device: Exablate 2100 — MRgFUS
  Arms: Treatment
Procedure: Myomectomy — Non-Hysteroscopic Myomectomy
  Arms: Surgery

SUMMARY:
The objective of this trial is to evaluate the safety and efficacy of ExAblate for the treatment of uterine fibroids.

Women, seeking treatment for symptomatic uterine leiomyomata will be eligible for the study.Women who agree to participate will sign an informed consent and will be randomized to ExAblate treatment or myomectomy.

All patients will be followed through the 36 month visit. Follow-up visits/telephone calls will be completed at 1 week, 2 weeks, 6 weeks, 3 months, 6, 12, 18, 24 and 36 months post treatment.

Patients will be evaluated by assessing their overall physical and mental health as well as for device/procedure related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18 or older
2. Symptomatic uterine fibroids, defined as those resulting in scores of 21 or higher, based on patient responses to questions 1-8 (raw score) of the Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire (UFS-QOL).
3. Women who have given written informed consent
4. Women who are able and willing to attend all study visits
5. Patient is pre or peri-menopausal (within 12 months of last menstrual period)
6. Able to communicate sensations during the ExAblate procedure
7. Uterine fibroids, which are device accessible
8. Fibroid(s) clearly visible on non-contrast MRI.
9. Fibroid(s) enhances on MR contrast imaging

Exclusion Criteria:

1. Women currently pregnant
2. Uterine size > 24 cm W/O the cervix
3. More than 4 clinically significant fibroids (per MRI)
4. Prior myomectomy, UAE
5. Allergy to either gadolinium or iodinated contrast
6. Implanted metallic device prohibiting MRI
7. Severe claustrophobia
8. Active pelvic infection
9. Current use of intrauterine contraceptive device
10. Unstable medical conditions requiring additional monitoring during the procedure
11. Bleeding diathesis requiring medical treatment
12. Imaging suggestive of malignant disease of uterus, ovary, or cervix
13. Imaging and suggestive of adenomyosis.
14. Pedunculated submucosal or pedunculated subserosal myoma
15. Size and weight which prohibits subject from fitting in MRI device
16. Unavoidable, scarring, skin folds or irregularity, bowel, pubic bone, IUD, surgical clips or hard implants in the beam path.
17. Hyper intense fibroid relatively to the uterus muscle
18. Women with ovarian dermoid cyst anywhere in the treatment path

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety | 36 months post treatment
  Safety will be evaluated by recording and assessing the incidence and severity of major adverse events from treatment through the 3 years follow-up period.
Efficacy | 36 months post treatment
  Comparison between ExAblate treatment and non-Hysteroscopic Myomectomy in terms of treated patients who did not undergo another interventional treatment for recurrence of uterine fibroid symptoms at up to 36 months (3 years).

SECONDARY OUTCOMES:
Efficacy | 36 months post treatment
  1. Post treatment change in patient's quality of life
  2. Post treatment change in pelvic pain
  3. Post treatment Change in bleeding
  4. Post treatment recovery time

CONTACTS AND LOCATIONS:
Overall Officials: Wady Gedroyc, Prof., Principal Investigator — St Mary's Hospital, London
Locations (1):
- St. Mary's Hospital, London, United Kingdom

REFERENCES:
- See also: Sponsor's website — http://www.insightec.com